CLINICAL TRIAL: NCT06841783
Title: Ultrasound-Guided Erector Spinae Plane Block Versus Modified Thoracoabdominal Nerve Block for Perioperative Analgesia in Obese Patients Undergoing Laparoscopic Sleeve Gastrectomy. A Randomized Comparative Trial
Brief Title: Ultrasound-Guided Erector Spinae Plane Block Versus Modified Thoracoabdominal Block for Analgesia in Obese Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Ahmed nabih youssef, lecturer of anesthesia, Kasr El Aini Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MS-375-2023
Record Dates: First submitted 2025-02-19; First posted 2025-02-24 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Obesity, Morbid
MeSH Terms: conditions — Obesity, Morbid | interventions — Nerve Block

STUDY DESIGN:
Intervention Model Description: Patients will be randomly allocated by a computer-generated table into two of the study groups, the randomization sequence had been concealed in sealed opaque envelopes that will be opened by third doctor who will not participating in the study. The details of the series will be unknown to the investigators and the group assignment will kept in a set of sealed envelopes each bearing only the case number on the outside.
  This study will be performed by 2 anesthetists; one anesthetist who is experienced in performing the blocks that allocated to perform either Erector Spinae block or modified thoracoabdominal nerve block.
  According to a computer-generated sequence of random numbers and sealed envelope, and the other anesthetist will be blinded to the technique performed, and will monitor the patients intra and postoperatively.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Erector Spinae Plane Block (Experimental): Ultrasound-Guided Erector Spinae Plane Block
  Interventions: Procedure: nerve block
- Modified Thoracoabdominal Nerve Block (Experimental): Ultrasound-Guided Modified Thoracoabdominal Nerve Block
  Interventions: Procedure: nerve block

INTERVENTIONS:
Procedure: nerve block — ultrasound guided nerve block

SUMMARY:
Obesity is a complex chronic disease that has become a major public health concern worldwide, with the prevalence of obesity increasing dramatically over the past few decades. Patients with morbid obesity pose a challenge for perioperative pain management. High ceiling analgesics-opioids have limited role due to safety concerns for patients with or without obstructive sleep apnea .

Insufficient postoperative pain management can have negative effects on recovery and quality of life, as well as limit patient comfort and delay the patient's ability to return to work after surgery .

Due to the numerous negative side effects of opioid drugs, including physical dependence, nausea, vomiting, and respiratory depression and subsequent airway obstruction, the Enhanced Recovery after Surgery (ERAS) guidelines for bariatric surgery currently advise opioid reduction in this procedure.

Ultrasound-guided erector spinae plane block (ESPB) and modified thoracoabdominal nerve block (M-TAPA) are both regional anesthesia techniques used to provide perioperative analgesia for obese patients undergoing LSG .

The ESPB targets the spinal nerves as they exit the erector spinae muscle, providing analgesia to the abdominal wall and paraspinal muscles. The technique has shown promising results in various surgical procedures and has a low risk of complications. By blocking the spinal nerves, the ESPB can provide effective pain relief in the postoperative period for patients undergoing LSG .

On the other hand, the M-TAPA targets the thoracic intercostal nerves and the abdominal wall, providing analgesia to these areas. The technique has been shown to provide effective perioperative analgesia in patients undergoing LSG. With or without ultrasound guidance, the use of M-TAPA can provide effective pain relief and reduce the need for opioid medication in the postoperative period.

This study aimed to compare the analgesic effect of ultrasound guided modified thoracoabdominal nerve block and an erector spinae plain block in patients undergoing LGS

DETAILED DESCRIPTION:
Patients will be randomly allocated into two groups: ESPB (n=20) and M TAPA (n=20).

1. ESPB group: This group will receive ultrasound guided erector spinae plane block.
2. M-TAPA group: This group will receive ultrasound guided modified thoracoabdominal nerve block.

Preoperative assessment:

The patient will enter the preparation room, he/she will be asked about his medical and surgical history in details and fasting hours (6-8 hrs) and full examination will be performed including airway examination. Lab investigations including complete blood count (CBC), coagulation profile, liver function tests and renal function tests will be checked.

The procedure will be explained to the patient and informed consent will be signed after his agreement then the patient will be classified into one of the groups.

The VAS will be explained to the patient in details as it will be used as a measurement tool for assessment of postoperative pain.

Operating Room preparation & Equipment:

The ultrasound used will be Siemens ACUSON X300 Ultrasound System, the scanning probe was a linear probe 8-14 MHZ. A 50-mm block needle 22 gauge will be used. (SonoPlex Stim Cannula, Germany) All blocks will be given by one researcher using 40ml of drug 0.25% bupivacaine (20ml on each side)

Intraoperative management:

After that, the patient will be monitored with electrocardiogram (ECG), non-invasive arterial blood pressure, pulse oximetry, oxygen saturation (SpO2) and Capnography. IV access will be secured with 18-gauge cannula and Premedication (ranitidine 2.0 mg/kg IV and metoclopramide 0.1 mg/kg IV) will be given. Predicted body weight will be used for calculation of drug dose.

A) In ESPB group:

* The patient will assume the sitting position with an assisting nurse for support and to ensure patient's safety.
* A single anesthesiologist will perform ESPB on both sides of the body.
* The level of T10 will be determined by counting 3 spinous processes below T7 (which is at the level of the inferior angle of the scapula), and will also be double-checked by counting down from C7.
* Before applying the block, the spinous process of the spine and a spot 3 cm laterally from it are indicated.
* The probe will then be lateralized 2.5-3 cm into the parasagittal plane.
* The needle will be placed and advanced under sono-vision until it contacts the transverse process of the T10 vertebra after being visible to the Trapezius, Rhomboid Major, Erector Spinae muscle, and these structures.
* No sedation will be used.
* Utilizing aseptic methods, subcutaneous local apathetic infiltration of lidocaine will be performed using insulin syringe.
* After negative aspiration, LA will be deposited deep to the erector spinae muscle in the fascial plane.
* After that, a 22-gauge spinal needle will be used to inject 20 ml of bupivacaine 0.25% and 5 ml of lidocaine 2% as local anesthesia (LA) on each side.

B) M TAPA group :

* The patient will assume the supine position with an assisting nurse for support and to ensure patient's safety.
* A single anesthesiologist will perform M-TAPA on both sides of the body.
* Transversus abdominis, internal oblique and external oblique muscles will be located with a high-frequency linear probe on the costochondral angle in the sagittal plane under ultrasound guidance at the 10th costal margin.
* In order to see the lower surface of the costal cartilage in the midline, a deep angle will be made to the costochondral angle at the margin of the 10th costa.
* Utilizing aseptic methods, subcutaneous local apathetic infiltration of lidocaine will be performed using insulin syringe.
* After negative aspiration, using the in-plane approach, a 22-gauge spinal needle will be placed in the cranial direction, and the needle's tip will then be advanced to the posterior aspect of the 10th costal cartilage.
* The 10th costal cartilage's cranial edge will be never passed by the needle tip, and 20 mL of 0.25% bupivacaine will be injected into the chondrium's lower surface.
* For the other side, the identical procedure will be repeated.

C) After blocks, the onset of general anesthesia will be achieved after intubation, surgical sterilization, draping and positioning.

D) All patients will receive general anaesthesia (GA). Anaesthesia will be induced with propofol (2 mg/kg), fentanyl (2 μg/kg) and atracurium (0.5 mg/kg). The GA will be maintained by isoflurane (1.2 %) and atracurium (0.1 mg/kg/20 min).

E) Intraoperative vital signs as heart rate, blood pressure and intraoperative opioid requirements will be recorded every 15 minutes till patient recovery.

F) After skin closure, muscle relaxation will be reversed using neostigmine (0.04mg/kg) and atropine (0.01mg/kg) after the return of spontaneous breathing.

G) Patients will be transferred to the post-anesthesia care unit (PACU) for 60 min for complete recovery and monitoring H) If at any point hypotension occurred (defined as a decrease in mean arterial pressure > 25% from the baseline value or systolic arterial pressure of 100 mmHg), it will be treated with 5 mg of IV bolus ephedrine, which will be repeated every 3 min until the hypotension resolved. Bradycardia (defined as a heart rate (HR) of 40 beats/min) will be treated with intravenous atropine (0.5 mg).

I) Within the first 30 minutes, postoperative vital signs (heart rate and blood pressure) and VAS (static and dynamic) for pain will be recorded at 30 minutes, 2, 6, 12, 24 hours and if VAS ≥4 or when the patient asks for analgesia, nalbuphine IV (0.1mg/kg) will be given (rescue analgesia) targeting VAS ≤ 3. The time to first call for analgesia will be recorded. The patient will receive paracetamol (1gm/8hrs IV) as a regular analgesia. If the patient requires more than two doses of rescue analgesia in the first hour following surgery, the block will be deemed to have failed. The inappropriate analgesia will be considered when 120% increase in systolic blood pressure and/or heart rate from baseline in absence of other causes. The intraoperative analgesic management will be achieved using fentanyl bolus of 1 mcg/kg.

ELIGIBILITY:
Inclusion Criteria:

* 1. ASA II & ASA III. 2. Gender both males and females 3. Age group: from 18 to 65 years old

Exclusion Criteria:

* • Patient refusal.

  * Uncooperative patients.
  * Allergy to local anesthetics.
  * Anatomical abnormality at injection site.
  * Redo or combined cholecystectomy surgery.
  * Infection at injection site.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2025-02-24 (Actual); Primary Completion 2026-01-06 (Actual); Study Completion 2026-01-06 (Actual)

PRIMARY OUTCOMES:
Time to first rescue analgesia | the first 24 hours postoperatively
  it is defined as time from extubation until time to first analgesic requirement during the first 24 hours postoperatively.

SECONDARY OUTCOMES:
The total opioid consumption | the first 24 hours postoperatively
  The total opioid consumption in mg

CONTACTS AND LOCATIONS:
Overall Officials: ahmed abdallah, Professor, Study Director — anesthesia department , cairo university
Locations (1):
- Kasr Alainy, Cairo, Egypt